CLINICAL TRIAL: NCT07272252
Title: Psychological Effects and Breastfeeding Self-Efficacy of a Structured Four-Step Narrative Nursing Intervention in Cesarean Mothers: A Randomized Controlled Mixed-Methods Study
Brief Title: Narrative Nursing for Cesarean Mothers' Anxiety and Breastfeeding Confidence
Acronym: NARRCARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xi Huang (Other)
Collaborators: Xiamen University (Other); Yilong People's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Xi Huang, Master's student, Xiamen University
Organization: Xiamen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: XMUNARRCARE2025; FJ2022B061 (Other Grant/Funding Number: Fujian Provincial Social Science Foundation); XMSHLXH2320 (Other Grant/Funding Number: Xiamen Nursing Association); Basic Nursing II (Other Grant/Funding Number: Fujian First-Class Undergraduate Program)
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Postpartum Anxiety; Postpartum Depression (PPD); Breastfeeding Self-Efficacy; Cesarean Section Wound
Keywords: narrative nursing; storytelling intervention; cesarean section; postpartum anxiety; breastfeeding confidence; mixed-methods; randomized controlled trial; China
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-center, two-arm, randomized, parallel-group, superiority trial with blinded outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine perinatal care (No Intervention): Participants receive standard ward education, nursing care, discharge instructions, and routine telephone follow-up without any additional narrative sessions.
- 4-step narrative nursing (Experimental): Participants receive usual care plus four nurse-led narrative sessions (pre-op externalization, post-op deconstruction, pre-discharge reconstruction, and 2-week meaning-reconstruction phone call) aimed at reducing anxiety and enhancing breastfeeding confidence.
  Interventions: Behavioral: 4-step narrative nursing program

INTERVENTIONS:
Behavioral: 4-step narrative nursing program — Four nurse-led storytelling sessions (pre-operative externalization, post-operative deconstruction, pre-discharge reconstruction, and 2-week meaning-reconstruction phone call) aimed at reducing anxiety and increasing breastfeeding self-efficacy.
  Arms: 4-step narrative nursing

SUMMARY:
This study tests whether a nurse-led "4-step narrative nursing" program can reduce anxiety and improve breastfeeding confidence in mothers who are having a planned or non-emergency cesarean section.

What is the problem? About 30-40% of Chinese cesarean mothers feel high anxiety after surgery, and 1 in 5 is at risk for postpartum depression. Low confidence in breastfeeding is also common.

What will we do?

We will randomly assign 160 mothers (1:1) to either:

Usual care - standard education and ward care, or

Usual care plus narrative nursing - four short (10-20 min) conversations with a trained nurse:

Before surgery - help the mother talk about her fears. 24-48 h after surgery - encourage her to "name" pain or worries and separate them from herself.

Before discharge - guide her to find positive moments and build a "strong-mom" story.

Two weeks later by phone - strengthen the new story and review feeding success. What will we measure? Main result: anxiety score at 48 h (STAI scale). Other results: depression risk, breastfeeding confidence, pain, and feeding rates up to 3 months.

Possible benefits:

Lower anxiety, better mood, higher breastfeeding rates. No drugs or extra procedures are involved, only talking.

Risks:

Minimal; some mothers may feel emotional during conversations, but nurses can pause or refer to counselling if needed.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-50 years
2. Scheduled for elective or non-emergency cesarean section at ≥37 weeks
3. Able to communicate in Mandarin and provide written informed consent
4. Expected hospital stay ≥24 h
5. Singleton pregnancy with stable maternal and neonatal condition allowing routine mother-baby contact

Exclusion Criteria:

1. Severe psychiatric disorders (schizophrenia, bipolar disorder, active suicidal ideation)
2. Maternal or neonatal need for ICU/NICU admission
3. Emergency cesarean section preventing baseline assessment
4. Communication or cognitive impairment precluding interview

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum anxiety at 48 hours | 48 hours post-surgery
  Mean score on the State-Trait Anxiety Inventory (STAI-State, 20 items) assessed 48 hours after cesarean delivery. Lower scores indicate less anxiety.

SECONDARY OUTCOMES:
Postpartum depression risk | 48 hours, 2 weeks, 3 months postpartum
  Proportion of women with Edinburgh Postnatal Depression Scale (EPDS) ≥ 10 at 48 hours, 2 weeks and 3 months.
Breastfeeding self-efficacy | 48 hours, 2 weeks, 3 months postpartum
  Mean score on the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF, 14 items) at 48 hours, 2 weeks and 3 months. Higher scores indicate greater confidence.
Pain intensity | 48 hours and 2 weeks postpartum
  Mean Numerical Rating Scale (NRS, 0-10) for self-reported pain at 48 hours and 2 weeks.
Breastfeeding continuation rate | 3 months postpartum
  Percentage of women who report any breastfeeding at 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Yilong County Maternal and Child Health Hospital, Nanchong, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Yes, we plan to share individual participant data (IPD). The de-identified IPD underlying published results will be made available to qualified researchers beginning 9 months after article publication and ending 36 months post-publication. Data access will be granted after approval of a methodologically sound proposal and execution of a data-sharing agreement. Interested parties should contact the corresponding author.
Supporting Information: Study Protocol, ICF
Time Frame: IPD and supporting information will be made available beginning 9 months after the primary results paper has been accepted for publication and ending 36 months after that date.
  An extension may be granted if a justifiable request is received before the closing date.
Access Criteria: Access is limited to qualified researchers with IRB/REC-approved, methodologically sound proposals relevant to the approved indication.
  Only de-identified participant data and the data dictionary will be provided. Requests should be e-mailed to 【corresponding-author@univ.edu】 with a 1-page protocol and statistical analysis plan.
  A data-sharing agreement outlining terms of use, confidentiality, and no attempt to re-identify participants must be signed before access is granted.
  Data will be shared through a password-protected secure cloud link; download is logged and audited.
URL: https://med.xmu.edu.cn/info/1055/2755.htm